CLINICAL TRIAL: NCT05347498
Title: Study on Efficacy and Safety of HR091506 Tablets in Treatment of Primary Gout With Hyperuricemia in Adults
Brief Title: A Trial of HR091506 Tablets in Treatment of Primary Gout With Hyperuricemia in Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR091506-103
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Primary Gout With Hyperuricemia in Adults
MeSH Terms: interventions — Febuxostat

STUDY DESIGN:
Intervention Model Description: HR091506 tablets compared with febuxostat tablets
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): HR091506 tablets + placebo of febuxostat tablets
  Interventions: Drug: HR091506 tablets + placebo of febuxostat tablets
- Treatment group B (Active Comparator): febuxostat tablets + placebo of HR091506 tablets
  Interventions: Drug: febuxostat tablets + placebo of HR091506 tablets

INTERVENTIONS:
Drug: HR091506 tablets + placebo of febuxostat tablets — HR091506 tablets 40mg qd + placebo of febuxostat tablets 40mg qd in Week 1 and 2, HR091506 tablets 80mg qd + placebo of febuxostat tablets 80mg qd in Week 3 and 4
  Arms: Treatment group A
Drug: febuxostat tablets + placebo of HR091506 tablets — febuxostat tablets 40mg qd + placebo of HR091506 tablets 40mg qd in Week 1 and 2, febuxostat tablets 80mg qd + placebo of HR091506 tablets 80mg qd in Week 3 and 4
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HR091506 tablets for treatment of primary gout with hyperuricemia in adults, and to compare the results with febuxostat tablets in the same doses.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years old, male or female.
2. BMI: 18.0 - 30 kg/m2.
3. Meet the 2015 ACR (American College of Rheumatology) gout classification criteria.
4. Fasting serum uric acid ≥480 μmol/L on 2 different days during the screening period.
5. Willing to use contraceptive measures during the study.
6. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. History of acute gout attack within 4 weeks before randomization.
2. Urinary calculi diagnosed by B-ultrasound within 4 weeks before randomization.
3. Subjects who have undergone major surgery or organ transplantation within 3 months before randomization.
4. Major cardiovascular disease within 6 months before randomization.
5. History of chronic infection or recurrent infection within 1 year before randomization.
6. History of malignant tumor or current history of combined malignant tumor within 5 years before screening.
7. History of secondary hyperuricemia, refractory gout, or xanthine metabolism disorder.
8. Subjects with poorly controlled blood pressure or diabetes mellitus.
9. History of chronic diffuse connective tissue disease and/or massively elevated urate diseases and/or untreated clinically significant thyroid disease.
10. History of diseases that may affect the in vivo process, safety evaluation, or subjects' participation in the research.
11. Abnormal laboratory tests that may affect subjects participating in the research.
12. Combined use of prohibited drugs.
13. Allergic to ingredient or component of the experimental drug.
14. Participated in other clinical trials within 1 month before randomization.
15. Pregnant or nursing women.
16. History of drug abuse, drug use and/or excessive drinking within 1 year before screening.
17. The inestigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with serum uric acid level < 360μmol/L on Day 15. | on Day 15.
Proportion of subjects with serum uric acid level < 360μmol/L at test of cure (TOC) | Test of cure, defined as the day after end of treatment, equivalent to Study Day 15 or 29

SECONDARY OUTCOMES:
The proportion of subjects with serum uric acid level < 300μmol/L on Day 15. | on Day 15.
Proportion of subjects with serum uric acid level < 360μmol/L at TOC | Test of cure, defined as the day after end of treatment, equivalent to Study Day 15 or 29
The proportion of subjects with serum uric acid level < 360μmol/L on Day 29. | on Day 29.
The proportion of subjects with serum uric acid level < 300μmol/L on Day 29. | on Day 29.
Change of serum uric acid level from baseline on Day 15 | from baseline on Day 15
Change of serum uric acid level from baseline on Day 29 | from baseline on Day 29

IPD SHARING:
Plan to Share IPD: Undecided